CLINICAL TRIAL: NCT05602792
Title: A Phase I/IIa Study to Assess the Safety, Tolerability, Biodistribution and Pharmacodynamic of T3011 Herpes Virus Administered Via Intratumoral Injection in Patients With Advanced Solid Tumors.
Brief Title: A Study of T3011 Administered Via Intratumoral Injection in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ImmVira Pharma Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TG1819ONC
Record Dates: First submitted 2022-10-18; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor; Sarcoma; HNSCC; Breast Cancer; Esophagus Cancer; NSCLC; Non-melanoma Skin Cancer
Keywords: Oncolytic virus; Herpes virus
MeSH Terms: conditions — Sarcoma; Squamous Cell Carcinoma of Head and Neck; Breast Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- T3011 Herpes Virus Injection (Experimental)
  Interventions: Biological: T3011

INTERVENTIONS:
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with advanced solid tumors.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with sarcoma.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with Malignant head and neck tumor.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with breast cancer.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with esophagus cancer.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with lung cancer.
Biological: T3011 — T3011 will be administered through intratumoral injection in patients with non-melanoma skin cancer.

SUMMARY:
A Phase I/IIa Study of the Safety and Tolerability of T3011 Administered via Intratumoral Injection in Patients with Advanced Solid Tumors

DETAILED DESCRIPTION:
This is a Phase I/IIa, open-label, first-in-human study of T3011 given via intratumoral (IT) injection in participants with advanced or metastatic solid tumors. Part I and part II of the study is a dose escalation which will use a 3+3 design to evaluate escalating doses of T3011. Part I is a single dose escalation. Part II is multiple dose escalation. Total enrollment will depend on the toxicities and/or activity observed, with approximately 8-48 evaluable participants enrolled.

Once the RP2D is established ,Part III will enroll approximately 40-60 participants with sarcoma , approximately 10-25 participants with Malignant head and neck tumor,approximately 10-25 participants with breast cancer,approximately 10-25 participants with esophagus cancer,approximately 10-25 participants with lung cancer and approximately 10-25 participants with non-melanoma skin cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age 18~70 years Part I ; Age 18 years or older (Part II and III ). 2. Histologically or pathologically confirmed diagnosis of locally recurrent or metastatic advanced malignancy.

  3. Measurable disease per RECIST version 1.1. 4. Must have at least 1 tumor lesion that is accessible for IT injection of T3011 in the opinion of the investigator.

  5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1. 6. Life expectancy > 12 weeks. 7. Women of child-bearing potential (WCBP) and men must agree to use adequate contraception prior to study entry, while on study treatment, and for six months after receiving last dose of T3011.

  8. WCBP must have a negative serum pregnancy test Within 7 days prior to W1D1. 9. Capable of understanding and complying with protocol requirements.

Exclusion Criteria:

* 1. Last dose of previous anticancer therapy < 4 weeks. 2. Prior treatment with another oncolytic virus or gene therapy. 3. Previous intolerance to anti-PD-(L)1 monoclonal antibody or previous history of immunotherapy induced non-infectious pneumonitis/interstitial lung disease.

  4. History of seizure disorders within 12 months of Screening. 5.History of allergic reactions attributed to compounds of similar biological composition to HSV-1, IL-12, or anti-PD-1 monoclonal antibody.

  6. Requires continued concurrent therapy with any drug active against HSV. 7. Pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Estimated)
Dates: Start 2020-04-21 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
In part I and part II, Evaluate the safety and tolerability of escalating doses of single dose and multiple dose IT T3011.Characterize DLTs and identify the MTD of IT T3011. | Up to 2 years from first dose of T3011
  Incidence rate of TEAE; Incidence rate of DLT
In part III, Evaluate the safety of multiple dose IT T3011 in the following indications,including sarcoma, Malignant head and neck tumor, breast cancer, esophagus cancer, lung cancer and non-melanoma skin cancer. | Up to 2 years from first dose of T3011
  Incidence rate of TEAE;

SECONDARY OUTCOMES:
In part I and part II, Characteristics of biological distribution and biological effect of single dose and multiple dose IT T3011. | Up to 2 years from first dose of T3011
  The changes of PD-1 and IL-12 concentration after administration
In part I and part II, Evaluation of pharmacodynamics of T3011 | Up to 2 years from first dose of T3011
  IFN-γ、 IL-1β、 IL-2、 IL-4、 IL-6、 IL-8、 IL-10、 IL-13、 TNF-α
In part I and part II, Evaluation of immunogenicity of T3011 | Up to 2 years from first dose of T3011
  ADAs and Nabs of IL-12, anti-PD-1 antibody and HSV-1
Overall response rate (ORR) | Up to 2 years from first dose of T3011
  ORR is defined as the proportion of participants who have a partial response (PR) or complete response (CR) to intervention, based on assessments by RECIST v1.1 and iRECIST.
Disease control rate (DCR) | Up to 2 years from first dose of T3011
  DCR is defined as the percentage of participants who have achieved CR, PR, or stable disease (SD) based on assessments by RECIST v1.1 and iRECIST.
Duration of response (DOR) | Up to 2 years from first dose of T3011
  DOR is defined as the time from the first met CR or PR until disease progression or death due to any cause, whichever occurs first.
Progression-free survival (PFS) | Up to 2 years from first dose of T3011
  PFS is defined as the time from enrollment to the first documentation of progressive disease (PD) or death from any cause, whichever occurs first per RECIST v1.1 and iRECIST.
In part III,Overall Survival (OS) | Up to 2 years from first dose of T3011
  OS is defined as the time from enrollment to death from any cause.

OTHER OUTCOMES:
In part II and part III,Exploring tumor immunomodulatory mechanism and histological changes after IT T3011 | Up to 2 months from first dose of T3011
  Assesse histological changes by immunohistochemical fluorescence detection
In part II and part III,Exploring the relationship between genetic changes and drug efficacy | Up to 2 months from first dose of T3011
  Genetic testing of tumor tissue
In part II and part III,Exploring the proliferation and activity of immune cells in blood after IT T3011 | Up to 2 years from first dose of T3011
  Analysis of immune cells in blood

CONTACTS AND LOCATIONS:
Locations (19):
- China (19):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The Fifth Affiliated Hospital of Sun Yat-sen University, Guanzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Zhejiang University Medical College, Hanzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hanzhou, Zhejiang
  - Peking University First Hospital, Beijing
  - Beijing Jishuitan Hospital, Beijing
  - Ninth People's Hospital,Shanghai Jiao Tong University School to Medicine, Shanghai
  - Fudan University Cancer Hospital, Shanghai
  - Zhongshan Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai
  - The Second People's Hospital of Shenzhen, Shenzhen

IPD SHARING:
Plan to Share IPD: Undecided